CLINICAL TRIAL: NCT00541463
Title: A Multicenter, Open-Label, Randomized, Study to Compare the Efficacy and Safety of Indinavir 800 mg b.i.d. Plus Ritonavir 100 mg b.i.d. Plus Two NRTIs vs. Nelfinavir 1250 mg b.i.d. Plus Two NRTIs in HIV-1 Seropositive Patients Who Have Failed or Are Intolerant to an NNRTI Containing Regimen
Brief Title: A Study of Indinavir Plus Ritonavir Plus Two NRTIs vs. Nelfinavir Plus Two NRTIs in HIV Positive Patients (0639-112)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0639-112; 2007_642
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: HIV Infections
Keywords: HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Duration of Therapy

INTERVENTIONS:
Drug: MK0639, indinavir sulfate / Duration of Treatment: 48 Weeks
Drug: Comparator: nelfinavir mesylate / Duration of Treatment: 48 Weeks

SUMMARY:
A study comparing Indinavir plus Ritonavir plus 2 NRTIs vs. Nelfinavir 1250 plus two nucleoside reverse transcriptase inhibitors (NRTIs) in the treatment of HIV positive patients who have not responded to or are intolerant to a non-nucleoside reverse transcriptase inhibitor (NNRTI) containing treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* HIV positive
* No active heart disease

Exclusion Criteria:

* Pregnant or breast feeding
* Unwilling to use birth control or abstinence to prevent pregnancy
* Received an investigational drug or vaccine within the past 30 days or is planning to receive other investigational study drug/vaccine or interferon while in the study
* Plan to receive NNRTIs while in the study
* Received therapy which lowers body's ability to fight infection within the past 30 days or while in the study
* Alcohol or substance abuse
* Hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2001-01; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Plasma viral RNA levels will be measured at predetermined time points to determine mean change

SECONDARY OUTCOMES:
CD4 cell counts will be measured at predetermined time points to determine change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html